CLINICAL TRIAL: NCT01783548
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, 12-Week, Clinical Study Designed to Assess the Efficacy and Safety of BDP Nasal Aerosol (80 mcg, Once Daily) in Pediatric Subjects (4 to 11 Years of Age) With PAR
Brief Title: Study of an Investigational Nasal Aerosol or Placebo in Children (Ages 4 to 11) With Perennial Allergic Rhinitis (PAR)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BDP-AR-306
Record Dates: First submitted 2013-01-31; First posted 2013-02-05 (Estimated); Results first posted 2015-10-12 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Allergic Rhinitis
Keywords: allergic rhinitis; pediatric subjects; BDP nasal aerosol
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BDP Nasal Aerosol 80 mcg/day (Experimental): BDP nasal aerosol: 80 mcg dose once daily in the morning. Participants/parents administer 40 mcg BDP (one spray per nostril) during the 12-week Treatment Period.
  Interventions: Drug: BDP Nasal Aerosol
- Placebo Nasal Aerosol (Placebo Comparator): Placebo nasal aerosol: Participants/parents administer placebo (no medication) (one spray per nostril) once daily in the morning during the 12-week Treatment Period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BDP Nasal Aerosol
  Other Names: Beclomethasone dipropionate; QNASL®
  Arms: BDP Nasal Aerosol 80 mcg/day
Drug: Placebo
  Arms: Placebo Nasal Aerosol

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Beclomethasone dipropionate (BDP) nasal aerosol in subjects with Perennial Allergic Rhinitis (PAR).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 4 to 11 years of age, inclusive, as of the Screening Visit (SV).
* A documented history of PAR to a relevant perennial allergen for a minimum of 12 months (6 months for subjects 4 to 5 years of age) immediately preceding the study Screening Visit (SV).
* A demonstrated sensitivity to at least one allergen known to induce PAR through a standard skin prick test.
* Other criteria apply.

Exclusion Criteria:

* History of physical findings of nasal pathology, including nasal polyps or other clinically significant respiratory tract malformations, recent nasal biopsy, nasal trauma (e.g., nasal piercing) or surgery, atrophic rhinitis, or rhinitis medicamentosa (all within the last 60 days prior to the Screening Visit [SV]).
* History of a respiratory infection or disorder (including, but not limited to bronchitis, pneumonia, chronic sinusitis or influenza) within the 14 days preceding the Screening Visit (SV), or development of a respiratory infection during the Run-In Period.
* Active asthma requiring treatment with inhaled or systemic corticosteroids and/or routine use of beta-agonists and any controller drug (e.g., theophylline, leukotriene antagonists). History of intermittent use (less than or equal to 3 uses per week) of inhaled short acting beta-agonists prior to the Screening Visit (SV) is acceptable.
* Have any of the following conditions that are judged by the investigator to be clinically significant and/or affect the subject's ability to participate in the clinical trial.
* Other criteria apply.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 547 (Actual)
Dates: Start 2013-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (63):
- United States (63):
  - Teva Investigational Site 10522, Hot Springs, Arkansas
  - Teva Investigational Site 10518, Costa Mesa, California
  - Teva Investigational Site 10526, Downey, California
  - Teva Investigational Site 10496, Huntington Beach, California
  - Teva Investigational Site 10536, Huntington Beach, California
  - Teva Investigational Site 10479, Mission Viejo, California
  - Teva Investigational Site 10524, Orange, California
  - Teva Investigational Site 10508, Paramount, California
  - Teva Investigational Site 10495, San Diego, California
  - Teva Investigational Site 10504, San Diego, California
  - Teva Investigational Site 10505, Stockton, California
  - Teva Investigational Site 10514, Centennial, Colorado
  - Teva Investigational Site 10503, Colorado Springs, Colorado
  - Teva Investigational Site 10499, Lawrenceville, Georgia
  - Teva Investigational Site 10474, Savannah, Georgia
  - Teva Investigational Site 10490, Stockbridge, Georgia
  - Teva Investigational Site 10498, Stockbridge, Georgia
  - Teva Investigational Site 10509, DeKalb, Illinois
  - Teva Investigational Site 10493, Normal, Illinois
  - Teva Investigational Site 10486, Indianapolis, Indiana
  - Teva Investigational Site 10494, Louisville, Kentucky
  - Teva Investigational Site 10515, North Dartmouth, Massachusetts
  - Teva Investigational Site 10540, Traverse City, Michigan
  - Teva Investigational Site 10513, Columbia, Missouri
  - Teva Investigational Site 10532, Missoula, Montana
  - Teva Investigational Site 10507, Brick, New Jersey
  - Teva Investigational Site 10534, Corning, New York
  - Teva Investigational Site 10492, Cortland, New York
  - Teva Investigational Site 10517, Niagara Falls, New York
  - Teva Investigational Site 10482, Rochester, New York
  - Teva Investigational Site 10535, Watertown, New York
  - Teva Investigational Site 10478, High Point, North Carolina
  - Teva Investigational Site 10516, Holly Springs, North Carolina
  - Teva Investigational Site 10485, Canton, Ohio
  - Teva Investigational Site 10480, Cincinnati, Ohio
  - Teva Investigational Site 10500, Cleveland, Ohio
  - Teva Investigational Site 10529, Middleburg Heights, Ohio
  - Teva Investigational Site 10537, Ashland, Oregon
  - Teva Investigational Site 10527, Medford, Oregon
  - Teva Investigational Site 10502, Portland, Oregon
  - Teva Investigational Site 10477, Blue Bell, Pennsylvania
  - Teva Investigational Site 10484, Upland, Pennsylvania
  - Teva Investigational Site 10511, Warwick, Rhode Island
  - Teva Investigational Site 10497, Charleston, South Carolina
  - Teva Investigational Site 10521, Orangeburg, South Carolina
  - Teva Investigational Site 10528, Knoxville, Tennessee
  - Teva Investigational Site 10483, Boerne, Texas
  - Teva Investigational Site 10489, Dallas, Texas
  - Teva Investigational Site 10520, Dallas, Texas
  - Teva Investigational Site 10476, El Paso, Texas
  - Teva Investigational Site 10491, Kerrville, Texas
  - Teva Investigational Site 10487, Plano, Texas
  - Teva Investigational Site 10501, Plano, Texas
  - Teva Investigational Site 10523, San Antonio, Texas
  - Teva Investigational Site 10531, San Antonio, Texas
  - Teva Investigational Site 10539, San Antonio, Texas
  - Teva Investigational Site 10475, Waco, Texas
  - Teva Investigational Site 10488, Salt Lake City, Utah
  - Teva Investigational Site 10506, Salt Lake City, Utah
  - Teva Investigational Site 10510, Salt Lake City, Utah
  - Teva Investigational Site 10519, Burke, Virginia
  - Teva Investigational Site 10481, Richmond, Virginia
  - Teva Investigational Site 10533, Richmond, Virginia

REFERENCES:
- [Derived] Berger WE, Jacobs RL, Amar NJ, Tantry SK, Li J, Small CJ. Efficacy and safety of beclomethasone dipropionate nasal aerosol in children with perennial allergic rhinitis. Ann Allergy Asthma Immunol. 2015 Aug;115(2):130-6. doi: 10.1016/j.anai.2015.05.012. Epub 2015 Jun 24. PMID 26115578

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 770 subjects were screened. The 547 participants were randomly assigned to either BDP nasal aerosol (80 mcg/day) or placebo nasal aerosol in a 2:1 ratio.
Period: Overall Study
Arm/Group | BDP Nasal Aerosol 80 mcg/Day | Placebo Nasal Aerosol
Started | 362 (Randomized) | 185 (Randomized)
Full Analysis Set (FAS) | 358 | 184
Completed | 328 | 167
Not Completed | 34 | 18
Not completed — Adverse Event | 8 | 4
Not completed — Withdrawal by Subject | 11 | 8
Not completed — Non-compliance | 4 | 0
Not completed — Protocol Violation | 2 | 2
Not completed — Lost to Follow-up | 8 | 3
Not completed — Lack of Efficacy | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat population which included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | BDP Nasal Aerosol 80 mcg/Day | Placebo Nasal Aerosol | Total
Number analyzed (Participants) | 362 | 185 | 547
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.0 (2.16) | 8.0 (2.23) | 8.0 (2.18)
Age, Customized [Number; unit: participants]
  4 to 5 years | 62 | 31 | 93
  6 to 11 years | 300 | 154 | 454
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 175 | 71 | 246
  Male | 187 | 114 | 301
Race/Ethnicity, Customized [Number; unit: participants]
  White | 272 | 145 | 417
  Black | 65 | 25 | 90
  Other | 25 | 15 | 40
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 144 | 75 | 219
  Not Hispanic or Latino | 217 | 110 | 327
  Unknown | 1 | 0 | 1
Weight [Mean (Standard Deviation); unit: kg] | 33.4 (13.40) | 33.8 (13.24) | 33.5 (13.34)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 18.6 (4.22) | 18.9 (4.33) | 18.7 (4.25)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Average Morning (AM) and Evening (PM) Subject-Reported Reflective Total Nasal Symptom Score (rTNSS) Over The First 6 Weeks Of Treatment In Subjects 6 To 11 Years Of Age
Description: Reflective TNSS is an evaluation of symptom severity over the past 12 hours prior to the recording of the score. Participants (with assistance from parents/guardians/caregivers, as needed) assessed and recorded four nasal symptoms (runny nose, nasal congestion, nasal itching, and sneezing) twice daily (AM and PM) using the following scale:
  * 0 = absent (no sign/symptom present)
  * 1 = mild (sign/symptom clearly present, but minimal awareness; easily tolerated)
  * 2 = moderate (definite awareness of sign/symptom that is bothersome but tolerable)
  * 3 = severe (sign/symptom that is hard to tolerate; causes interference with activities of daily living and/or sleeping) The total TNSS scale was 0-12 with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms.
  Baseline and the during study rTNSS values were defined as the average AM and PM subject-reported rTNSS during each time period.
Time Frame: Baseline (Day -4 to Day 1 predose), Day 1 (postdose) to Week 6
Population: Full analysis set (FAS) included all participants in the ITT population who received at least 1 dose of randomized study medication and had at least 1 post-baseline subject-reported rTNSS assessment. Subpopulation of study participants aged 6-11 years.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BDP Nasal Aerosol 80 mcg/Day | Placebo Nasal Aerosol
Number analyzed (Participants) | 296 | 153
units on a scale | -2.26 (0.12) | -1.60 (0.17)
Statistical Analysis 1: Comparison: BDP Nasal Aerosol 80 mcg/Day vs Placebo Nasal Aerosol; Based on other studies, the standard deviation for the change from baseline over the first 6 weeks of treatment in the average of AM and PM rTNSS is assumed to be 2.0. Using this standard deviation, 450 subjects aged 6 to 11 years (300 on active treatment of BDP and 150 on placebo) provide approximately 90% power to detect a difference of 0.65 in rTNSS change from baseline between treatment groups with a two-sided alpha level of 0.05; Test type: Superiority or Other; p = 0.002, mixed-model for repeated measures (MMRM) — a priori statistical significance is <0.05; The MMRM included covariate adjustment for baseline, day, treatment, and the treatment by day interaction; LSM treatment difference from placebo = -0.66, 95% CI 2-sided [-1.08 to -0.24]

2. Secondary Outcome: Change From Baseline in the Average Morning (AM) and Evening (PM) Subject-Reported Instantaneous Total Nasal Symptom Score (iTNSS) Over The First 6 Weeks Of Treatment In Subjects 6 To 11 Years Of Age
Description: Instantaneous TNSS is an evaluation of symptom severity over the last 10 minutes prior to the recording of the score. Participants (with assistance from parents/guardians/caregivers, as needed) assessed and recorded four nasal symptoms (runny nose, nasal congestion, nasal itching, and sneezing) twice daily (AM and PM) using the following scale:
  * 0 = absent (no sign/symptom present)
  * 1 = mild (sign/symptom clearly present, but minimal awareness; easily tolerated)
  * 2 = moderate (definite awareness of sign/symptom that is bothersome but tolerable)
  * 3 = severe (sign/symptom that is hard to tolerate; causes interference with activities of daily living and/or sleeping) The total TNSS scale was 0-12 with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms.
  Baseline and the during study iTNSS values were defined as the average AM and PM subject-reported iTNSS during each time period.
Time Frame: Baseline (Day -4 to Day 1 predose), Days 1 (postdose) to Week 6
Population: Full analysis set (FAS). Subpopulation of study participants aged 6-11 years.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BDP Nasal Aerosol 80 mcg/Day | Placebo Nasal Aerosol
Number analyzed (Participants) | 296 | 153
units on a scale | -1.98 (0.12) | -1.39 (0.17)
Statistical Analysis 1: Comparison: BDP Nasal Aerosol 80 mcg/Day vs Placebo Nasal Aerosol; Test type: Superiority or Other; p = 0.004, mixed-model for repeated measures (MMRM) — a priori statistical significance is <0.05; The MMRM included covariate adjustment for baseline, day, treatment, and the treatment by day interaction; LSM treatment difference from placebo = -0.58, 95% CI 2-sided [-0.99 to -0.18]

3. Secondary Outcome: Change From Baseline in the Average Morning (AM) and Evening (PM) Subject-Reported Reflective Total Nasal Symptom Score (rTNSS) Over The First 6 Weeks Of Treatment In Subjects 4 To 11 Years Of Age
Description: as for outcome 1
Time Frame: Baseline (Day -4 to Day 1 predose), Day 1 (postdose) to Week 6
Population: Full analysis set (FAS) included all participants in the ITT population who received at least 1 dose of randomized study medication and had at least 1 post-baseline subject-reported rTNSS assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BDP Nasal Aerosol 80 mcg/Day | Placebo Nasal Aerosol
Number analyzed (Participants) | 358 | 184
units on a scale | -2.32 (0.11) | -1.71 (0.16)
Statistical Analysis 1: Comparison: BDP Nasal Aerosol 80 mcg/Day vs Placebo Nasal Aerosol; Test type: Superiority or Other; p = 0.002, mixed-model for repeated measures (MMRM) — a priori statistical significance is <0.05; The MMRM included covariate adjustment for baseline, day, treatment, and the treatment by day interaction; LSM treatment difference from placebo = -0.62, 95% CI 2-sided [-1.00 to -0.23]

4. Secondary Outcome: Change From Baseline in the Average Morning (AM) and Evening (PM) Subject-Reported Instantaneous Total Nasal Symptom Score (iTNSS) Over The First 6 Weeks Of Treatment In Subjects 4 To 11 Years Of Age
Description: as for outcome 2
Time Frame: Baseline (Day -4 to Day 1 predose), Days 1 (postdose) to Week 6
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BDP Nasal Aerosol 80 mcg/Day | Placebo Nasal Aerosol
Number analyzed (Participants) | 358 | 184
units on a scale | -2.07 (0.11) | -1.53 (0.15)
Statistical Analysis 1: Comparison: BDP Nasal Aerosol 80 mcg/Day vs Placebo Nasal Aerosol; Test type: Superiority or Other; p = 0.004, mixed-model for repeated measures (MMRM) — a priori statistical significance is <0.05; The MMRM included covariate adjustment for baseline, day, treatment, and the treatment by day interaction; LSM treatment difference from placebo = -0.54, 95% CI 2-sided [-0.91 to -0.17]

ADVERSE EVENTS:
Time Frame: Day 1 to Week 16
Arm/Group | BDP Nasal Aerosol 80 mcg/Day | Placebo Nasal Aerosol
Serious Adverse Events (participants affected / at risk) | 0/362 | 0/185
Other Adverse Events (participants affected / at risk) | 33/362 | 21/185
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BDP Nasal Aerosol 80 mcg/Day (N=362) | Placebo Nasal Aerosol (N=185)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 18 | 8
Headache (Nervous system disorders) | 16 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.